CLINICAL TRIAL: NCT00674427
Title: A Phase I/II Trial Of DLI And Activated DLI (ADLI) Followed By Either Repetitive Dosing Of ADLI Or Dose Escalated ADLI For Patients With Relapse After Allogeneic Stem Cell Transplantation
Brief Title: Trial of Donor Lymphocyte Infusion (DLI) and Activated DLI Following Relapse After Allogeneic Stem Cell Transplant
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient funds
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 805534 UPCC 20406
Record Dates: First submitted 2008-05-05; First posted 2008-05-07 (Estimated); Last update posted 2020-08-17 (Actual); Status verified 2020-08

CONDITIONS: Chronic Myelogenous Leukemia; Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndrome; Non-Hodgkin's Lymphoma; Hodgkin's Disease; Multiple Myeloma; Chronic Lymphocytic Leukemia
Keywords: AML; ALL; MDS; CLL; Multiple Myeloma
MeSH Terms: conditions — Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CR (Experimental): Subjects who are in CR ater 6-12 weeks after aDLI
  Interventions: Biological: CD3/CD28 Activated T cells
- Not in CR (Experimental): Subjects not in CR after 6-12 weeks after aDLI
  Interventions: Biological: CD3/CD28 Activated T cells

INTERVENTIONS:
Biological: CD3/CD28 Activated T cells — Subjects who are not in CR will receive one infusion of high dose aDLI
  Arms: Not in CR
Biological: CD3/CD28 Activated T cells — Subjects in CR 6-12 weeks after the first dose of Activated Donor Lymphocyte Infusion (aDLI) will continue to receive aDLI every 3 months for up to a year.
  Arms: CR

SUMMARY:
This study is for patients with relapsed of disease after allogeneic bone marrow

The donor's T cells are activated by exposure to 2 compounds or antibodies that bind (or stick to) two compounds on T cells called CD3 and CD28. When these antibodies stick to both CD3 and CD28 on the T cells, the T cells becomes stimulated (or "activated") and grows. CD3 and CD28 are the coating of a T cell and a T cell is part of the body's immune system.

It is believed that when T cells are exposed to both of antibodies to CD3 and CD28 compounds at the same time, they become activated or "stimulated" and may be more effective in fighting infections or cancer cells. We call this therapy "activated donor lymphocyte infusions, or activated DLI (aDLI)".

This current study is being performed to see whether it is safe and effective to administer higher doses of activated DLI or repeated doses of activated DLI.

All patients will receive standard donor lymphocyte infusions first, and in addition will receive activated donor lymphocytes approximately 12 days later (DLI followed by aDLI). Depending on the response to this treatment, and depending on possible side effects (such as graft-vs-host disease as described below), patients in remission will then receive additional aDLI every 3 months for 4 more times, and patients not in remission within 6-12 weeks will receive higher dose aDLI. The timing of the higher dose aDLI will be determined by your physician depending on your disease and the rate of progression of your disease. The aDLI can be given as early as 6 weeks, or as late as 12 weeks (3 months).

DETAILED DESCRIPTION:
You are being asked to participate in this research study because your disease has relapsed after allogeneic bone marrow transplantation (putting normal bone marrow from one person into another that was a brother/sister, a matched family member, or an unrelated donor). This study is testing a treatment for your relapsed disease after bone marrow transplant (BMT) that uses infusions of your bone marrow donor's immune cells (system which protects the body from disease); these immune cells are white blood cells called leukocytes or lymphocytes (called T cells). In allogeneic BMT, we know that the donor's immune system (system which protects the body from disease and is comprised primarily of lymphocytes, or white blood cells) is very important for the control and elimination of leukemia after bone marrow transplantation. Many studies have shown that treatment with transfusions of the bone marrow donor's lymphocytes can lead to a complete remission in patients that have relapsed after BMT. This procedure is called donor lymphocyte infusion, or "DLI". The conventional or standard way to give donor lymphocyte infusions (referred to as DLI) is to take the lymphocytes from the blood of the original bone marrow donor blood and infuse them directly into a patient with relapsed disease without any processing of the lymphocytes.

Some patients have a very good chance of achieving remission after donor lymphocyte infusions (such as patients with early stages of CML). Standard DLI after allogeneic BMT have been less effective for patients with advanced leukemia (AML, ALL, or "accelerated phase" and "blast crisis" CML), or patients with other diseases such as myelodysplasia, CLL, Hodgkin's lymphoma and non-Hodgkin's lymphoma. Because of your disease, your physician estimates a chance of less than 4 in 10 (40%) or less of responding to standard donor lymphocyte infusions (DLI).

In a recent clinical trial, we tested the safety of a new way to give DLI that might make this treatment more effective. The donor lymphocytes (or T cells) are activated in the laboratory before given to patients to try and make them more active. The donor's T cells are activated by exposure to 2 compounds or antibodies that bind (or stick to) two compounds on T cells called CD3 and CD28. When these antibodies stick to both CD3 and CD28 on the T cells, the T cells becomes stimulated (or "activated") and grows. CD3 and CD28 are the coating of a T cell and a T cell is part of the body's immune system.

It is believed that when T cells are exposed to both of antibodies to CD3 and CD28 compounds at the same time, they become activated or "stimulated" and may be more effective in fighting infections or cancer cells. We call this therapy "activated donor lymphocyte infusions, or activated DLI (aDLI)".

In a previous study in which patients received standard DLI and aDLI, we felt that responses were at least as good as conventional DLI but too few patients were treated to know if responses might be better. Unfortunately, as noted in other studies using DLI, about half of the patients did not respond, and about half of the patients in remission had later relapse of their disease.

This current study is being performed to see whether it is safe and effective to administer higher doses of activated DLI or repeated doses of activated DLI.

* Patients who are in remission at 3 months after receiving the initial activated DLI will be treated with more activated donor lymphocytes every 3 months for a total of 4 more times (3 months, 6 months, 9 months and 12 months after the first infusion) to test if it is safe to give repeated doses of activated DLI and to see if repeated doses will prevent subsequent relapse.
* For those patients who are not in remission 6-12 weeks after the initial activated DLI, we will test whether it is safe and effective to give higher doses of activated donor lymphocytes. Using the experimental procedures that activate the donor lymphocytes, lymphocytes can also be grown up in the laboratory and 10 times more lymphocytes can be given to you than can be obtained using more conventional DLI.

For this study, similar to our previous study with aDLI, all patients will receive standard donor lymphocyte infusions first, and in addition will receive activated donor lymphocytes approximately 12 days later (DLI followed by aDLI). Depending of the response to this treatment, and depending on possible side effects (such as graft-vs-host disease as described below), patients in remission will then receive additional aDLI every 3 months for 4 more times, and patients not in remission within 6-12 weeks will receive higher dose aDLI. The timing of the higher dose aDLI will be determined by your physician depending on your disease and the rate of progression of your disease. The aDLI can be given as early as 6 weeks, or as late as 12 weeks (3 months).

In the previous study the highest dose of aDLI a patient received is the same as the dose to be initially administered in this study which is 1 x 108 CD3+ cells/kg. However, this research study will also include doses higher than those used in the previous study. Patients in remission will receive the same dose of 1 x 108 CD3+ cells/kg on 4 additional occasions as long as no unacceptable side effects are observed. Patients that are not in remission will receive a dose that is 10 times higher.

ELIGIBILITY:
Inclusion Criteria:

* Prior allogeneic stem cell transplant.
* Expected survival > 4 weeks
* Original bone marrow donor available for leukocyte donation.
* Absence of active acute GVHD > grade I, or chronic GVHD.
* Off all immune suppression for GVHD for 28 days (an exception may be made for patients with acute leukemia whose disease is progressing rapidly and a 28 day waiting period after discontinuation of immune suppression is not practical or appropriate).
* Creatinine < 2.5 mg/dl.
* Relapsed or persistent advanced malignancy with less than a 50% chance of responding to unstimulated DLI:

  a. CML: Relapse with accelerated phase, or blast phase disease b. AML, ALL i. Cytogenetic relapse (less than 5% blasts).
  1. The patient's leukemia-specific chromosome abnormality is detectable by standard cytogenetics in more than 25% of cells at any time greater than day 50 post-transplant.

     ii. Hematologic relapse: More than 5% blasts in the marrow or peripheral blood.

     c. MDS d. Non-Hodgkin's Lymphoma or Hodgkin's Disease i. Relapse: Recurrent disease by serial physical exam, radiographic studies, or molecular studies. If possible, tumor should be re-biopsied to determine histology and rule out possibility of EBV-related lymphoproliferative disease e. CLL f. Myeloma

     Exclusion Criteria:
* Active chronic or acute GVHD > grade I.
* Requirement for active immunosuppression to treat GVHD.
* Pregnant or lactating women. The safety of this therapy on unborn children or effects on breast milk are not known.
* Uncontrolled active infection
* Any uncontrolled active medical disorder that would preclude participation as outlined.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2008-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Determining the incidence and severity of acute and chronic GVHD associated with repetitive dosing of aDLI. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: David Porter, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No